CLINICAL TRIAL: NCT06886152
Title: Transcutaneous Spinal Stimulation and Gait Training to Improve Mobility and Motor Control in Individuals With Traumatic Brain Injury
Brief Title: Spinal Stimulation and Gait Training to Improve Mobility in TBI
Acronym: DOD SS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Karen J. Nolan, PhD, Associate Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1260-24
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; Traumatic Brain Injury (TBI); Hemiplegia and Hemiparesis
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemiplegia; Paresis | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TBI with Stim (Experimental): Participants with TBI will be asked to come in 3 days a week for 6 weeks for walking training provided by a trained, licensed physical therapist. Electrodes will be placed on the surface of the skin along the spinal cord to provide stimulation during walking.
  Interventions: Procedure: Transcutaneous Spinal Cord Stimulation
- TBI with Sham (Sham Comparator): Participants with TBI will be asked to come in 3 days a week for 6 weeks for walking training provided by a trained, licensed physical therapist. Electrodes will be placed on the surface of the skin along the spinal cord but will not provide stimulation during walking.
  Interventions: Other: Sham

INTERVENTIONS:
Procedure: Transcutaneous Spinal Cord Stimulation — A portable transcutaneous spine stimulator (Digitimer ®, USA) will supply biphasic stimulation superficial to the thoracolumbar spine.
  Arms: TBI with Stim
Other: Sham — A portable transcutaneous spine stimulator (Digitimer ®, USA) will be applied superficially with no electrical current.
  Arms: TBI with Sham

SUMMARY:
The purpose of this research study is to assess the effects of receiving transcutaneous spinal stimulation while performing walking exercises compared to completing walking exercises without spinal stimulation for individuals with hemiplegic TBI.

DETAILED DESCRIPTION:
The fundamental hypothesis guiding this proposal is that transcutaneous spinal cord stimulation combined with gait training for individuals with hemiplegic TBI will lead to improved: modulation of corticospinal networks, functional mobility, gait symmetry, standing posture, balance, and motor efficiency compared to gait training with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Have weakness on at least one side of my body.
* No injury to my unaffected side in 6 months.
* Be cleared by a physician to participate in this study.
* Have had a non-penetrating TBI at least 2 years ago. A non-penetrating injury is an injury where my skull remained closed and no object entered it.
* Have enough strength to use a hemiwalker or walker.
* Be between 18-65 years of age.
* Be medically stable for at least 6 months before enrolling. This means that I have not had an emergency room visit, hospitalization, or medical procedure (such as a surgery) during this period of time.
* Able to walk 10 yards with minimal assistance without an ankle-foot orthosis (brace)
* Able to respond to and tolerate surface stimulation, as determined by study staff
* Have the ability to communicate in English.
* Have stable blood pressure.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, verbal instructions, and follow-up requirements.

Exclusion Criteria:

* Have must have not had physical or occupational therapy or treatment for a balance disorder within 30 days prior to study enrollment. I must not participate in physical or occupation therapy throughout the duration of the study to avoid affecting the study results.
* Have any medical issues that affect my unaffected side (such arthritis, fracture, etc.).
* Have skin issues that would prevent me from being able to use the surface stimulation (such as a open wound or rash).
* Have a pre-existing condition that may make it difficult for me to participate in exercise. (uncontrolled hypertension as described by a physician, heart disease, abnormal heart rate or rhythm, or congestive heart failure).
* Have been hospitalized for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Have an implanted medical or metallic device.
* Reduced sensation in my lower limbs and stimulation locations.
* Have Botox injections in my legs up to 3 months prior to enrolling.
* Have physical therapy for walking.
* Have uncontrolled seizure disorder (such as epilepsy)
* Have nervous system-related issues (for example Parkinson's disease, multiple sclerosis).
* Major changes to my medications throughout the study
* Have bone or muscle issues unrelated to traumatic brain injury that interfere with my walking or limit my range of motion in my legs.
* Be currently pregnant. Because of potential risk to the fetus, women of child bearing potential will be required to have a pregnancy test before they can enroll in this study. If I am female, and have a positive pregnancy test, I will not be enrolled.
* Have any other medical conditions that my doctor or physical therapist feels would affect my ability to use the stimulation or participate in walking training TMS Specific - Exclusion (those with these exclusions can still participate in other parts of the study)
* I have a history of seizure disorder or have a close family member (parent, brother, sister, or child) who has a seizure disorder.
* I have had unexplained fainting spells.
* I have had an active migraine headaches.
* I have a past or current history of ringing in the ears (tinnitus) or severe hearing problems.
* I am currently taking or withdrawing from any medication that would increase my risk of seizure (determination made in consultation with study physician).
* I have a history of alcohol or drug abuse in the prior 3 years.
* I have nerve damage outside of my brain or spinal cord (such as in an arm or leg).
* I am unwilling to participate in TMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
10MWT (Aim 1) | Change from Baseline 10MWT at 6 weeks and 3 months
  10 meter walk test is a timed test to evaluate walking speed after TBI and in response to the intervention.
6MWT (Aim 1) | Change from Baseline 6MWT at 6 weeks and 3 months
  6 minute walking test to evaluate endurance after TBI and in response to the intervention. Distance is measured for 6 minutes with a greater distance indicating a better outcome.
TUG (Aim 1) | Change from Baseline 6MWT at 6 weeks and 3 months
  Timed up and go (TUG) is a timed test to measure functional balance and walking ability after TBI and in response to the intervention.
DGI (Aim 1) | Change from Baseline DGI at 6 weeks and 3 months
  Dynamic Gait Index (DGI) evaluates the ability to modify balance while walking in the presence of external demands after TBI and in response to the intervention. The measure is scored out of 24 with a higher score indicating a better outcome.
Berg Balance Scale (Aim 1) | Change from Baseline Berg at 6 weeks and 3 months
  Measure to assess static and dynamic balance and fall risk after TBI and in response to the intervention. The scale is scored out of 56 with a high score indicating a better outcome.
Temporospatial Loading (Aim 1) | Change from Baseline at 6 weeks and 3 months
  Step length, timing during gait cycle, limb symmetry will be collected using instrumented gait walkway and are combined to evaluate gait symmetry.
Joint Range of Motion (kinematics) (Aim 2) | Change from Baseline at 6 weeks and 3 months
  Kinematics gait data will be collected using a motion capture camera system to provide biomechanical outcomes.
Transcranial magnetic stimulation (TMS) (Aim 2) | Change from Baseline at 6 weeks and 3 months
  Transcranial magnetic stimulation (TMS) will be used to assay changes in cortical neurophysiology for all subjects using Magstim Rapid2TM 70 mm double coil (or similar device).
Participation Objective Participation Subjective (Aim 3) | Change from Baseline at 6 weeks and 3 months
  The POPS consists of 26 elements of participation representing 5 categories. For each item the participant rates each element objectively and subjectively.
Community Integration Questionnaire (Aim 3) | Change from Baseline at 6 weeks and 3 months
  The CIQ is a 15-item instrument used to assess the social role limitations and community interaction of people with brain injury with higher scores indicating greater independence and community integration.
Patient Competency Rating Scale (Aim 3) | Change from Baseline at 6 weeks and 3 months
  The PCRS is a 30 item self report scale using a 5 point Likert to rate the degree of difficulty in a variety of tasks and functions including measure of awareness of deficits following TBI in daily living, behavioral and emotional function, cognitive abilities, and physical function. Higher score indicates greater competency.
Perceived Control Scale for Brain Injury (Aim 3) | Change from Baseline at 6 weeks and 3 months
  This scale is 9 items scored on a 4 point Likert. It measures perceived control developed for individuals with acquired brain injury with a higher score indicating higher perceived control.
SF-36 (Aim 3) | Change from Baseline at 6 weeks and 3 months
  The Short Form (SF) Survey is the most widely used and studied measure of health-related quality of life consisting of 36 items, completed by the participant. Higher average scores indicate a more favorable state of health.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: No